CLINICAL TRIAL: NCT00509678
Title: Phase IB, Investigator-Initiated, Open-Label, Multi-Center Trial of Rituximab With or Without Methotrexate In Subjects With Psoriatic Arthritis and Psoriasis
Brief Title: Rituxan With or Without Methotrexate in Psoriatic Arthritis
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Swedish Medical Center (Other)
Collaborators: Genentech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: U3081n
Record Dates: First submitted 2007-07-27; First posted 2007-07-31 (Estimated); Last update posted 2012-01-18 (Estimated); Status verified 2012-01

CONDITIONS: Psoriatic Arthritis
Keywords: Rituximab; Rituxan; Psoriatic Arthritis; Arthritis
MeSH Terms: conditions — Arthritis, Psoriatic; Arthritis | interventions — Rituximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: Rituximab — 1000mg (1gm) given as an IV infusion every two weeks for 2 doses (days 1 and 15). The first infusion of rituximab should be administered IV at an initial rate of 50 mg/hr. If a hypersensitivity or infusion related reaction does not occur, escalate the infusion rate by 50 mg/hr increments every 30 minutes, to a maximum of 400 mg/hr.
  Other Names: Rituxan

SUMMARY:
The purpose of this study is to help determine the effectiveness of rituxan (with or without methotrexate) in the treatment of psoriatic arthritis.

DETAILED DESCRIPTION:
The purpose of this study is to evaluate safety and efficacy of rituximab, with and without methotrexate, in joints, enthesium and skin in psoriatic arthritis patients with inadequate response to methotrexate who have either not tried anti-TNF therapy or have had inadequate or failed response to anti-TNF therapy. To explore biologic mechanism of action via histological and immunohistochemical evaluation of pre and post treatment biopsies of psoriatic plaques.

ELIGIBILITY:
Inclusion Criteria:

* Active disease of at least 6 months duration.
* Receiving treatment on an outpatient basis.
* The patient will have at least one evaluable skin plaque, 2 cm in diameter, that can be followed with a target lesion score (scalp and groin lesions cannot be used).
* Presence of PsA per the CASPAR categories: Psoriasis, Nail Changes, Negative RF test, Dactylitis or radiological evidence of juxta-articular new bone formation.
* Subjects will have greater than or equal to 3 tender (out of 68 joints) and 3 swollen (out of 66) joints at screening and baseline.

Exclusion Criteria:

* History of malignancy other than resolved squamous or basal cell or cervical carcinoma
* Presence of a significant medical illness that, in the opinion of the investigator, would potentially compromise the subject's ability to participate in the trial
* Presence of another rheumatic or skin disease that, in the opinion of the investigator, could confound the ability to discern response
* History or presence of HIV
* History of severe allergic or anaphylactic reactions to humanized or murine monoclonal antibodies
* History of recurrent significant infection or history of recurrent bacterial infections
* Known active bacterial, viral, fungal, mycobacterial, or other infection (including tuberculosis or atypical mycobacterial disease, but excluding fungal infections of nail beds) or any major episode of infection requiring hospitalization or treatment with i.v. antibiotics within 4 weeks of screening or oral antibiotics within 2 weeks prior to screening.
* History of psychiatric disorder that, in the judgment of the investigator, would make the patient inappropriate for entry into this trial or would lead to poor compliance.
* Concurrent treatment with any DMARD (except for MTX), any anti-TNF alpha therapy or other biologic therapy. Topical medications to treat psoriasis are limited to class VI and VII low potency steroids to the palms, soles of the feet, axilla and groin only.
* Concurrent treatment with any DMARD (except for MTX), any anti-TNF alpha therapy or other biologic therapy. Topical medications to treat psoriasis are limited to class VI and VII low potency steroids to the palms, soles of the feet, axilla and groin only.
* Treatment with any investigational agent within 4 weeks of screening or 5 half-lives of the investigational drug (whichever is longer).
* Previous treatment with any cell-depleting therapies, including investigational agents (e.g., CAMPATH, anti-CD4, anti-CD5, anti-CD3, anti-CD19).
* Previous treatment within 6 months with i.v. gamma-globulin, Orencia, toclizumab, natalizumab or Prosorba Column.
* Intra-articular or parental corticosteroid injections within 4 weeks prior to screening.
* Previous treatment with rituximab (MabThera/Rituxan)
* Immunization with a vaccine within 4 weeks prior to randomization (e.g.; MMR, Varivax, Smallpox).
* One intra-articular steroid joint injection is allowed, affected joint is excluded from assessment thereafter.
* Subjects should not take analgesics within 12 hours prior to joint assessments

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2006-12; Primary Completion 2010-01 (Actual); Study Completion 2010-03 (Actual)

PRIMARY OUTCOMES:
Safety of Rituximab in PSA and psoriasis by determining incidence of treatment emergent AE's including infections, infusion reactions and disease progression. | followed out for one year from last dose

SECONDARY OUTCOMES:
The exploration of efficacy of rituximab in PsA will be determined by using the week 24 ACR 20 measurement as modified for PsA using 68/66 tender/swollen joint count. | Week 24

CONTACTS AND LOCATIONS:
Overall Officials: Philip J Mease, MD, Principal Investigator — Seattle Rheumatology Associates/ Swedish Research Center
Locations (4):
- United States (4):
  - University of California, San Diego, La Jolla, California
  - Stanford University, Stanford, California
  - University of Rochester, Rochester, New York
  - Swedish Rheumatology Research, Seattle, Washington